CLINICAL TRIAL: NCT03760120
Title: Short-term Effects of Positive Expiratory Pressure Mask on Ventilation Inhomogeneity in Children and Adolescents With Cystic Fibrosis
Brief Title: Short-term Effects of Physiotherapy on LCI
Acronym: SPICy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2291
Record Dates: First submitted 2018-11-07; First posted 2018-11-30 (Actual); Last update posted 2022-12-29 (Actual); Status verified 2022-12

CONDITIONS: Cystic Fibrosis
Keywords: physiotherapy; pulmonary function
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Intervention Model Description: Cross-over randomized controlled trial. Procedure: two nitrogen multiple-breath washout tests, one before and one after the intervention with PEP-Mask, either standard or sham allocation, during two subsequent mornings.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Technicians performing multiple-breath washout tests are blinded to treatment allocation; physiotherapists performing the treatment are blinded to multiple breath washout results; patients are blinded to the purpose of the study; the statistician will be blind to treatment allocation together with outcome assessors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEP standard (Active Comparator)
  Interventions: Device: PEP-MASK
- PEP sham (Sham Comparator)
  Interventions: Device: PEP-MASK

INTERVENTIONS:
Device: PEP-MASK

SUMMARY:
Although some studies have brought some evidences about the efficacy of positive expiratory pressure (PEP)-mask therapy as an airway clearance technique, yet it is not clearly understood what is the contribution of this technique in modifying peripheral ventilation inhomogeneity, a typical feature of patients with Cystic Fibrosis (CF).

The aim of this study is to investigate how PEP-MASK affects ventilation inhomogeneity in children and adolescents, with moderate to normal CF lung disease by the change in acinar airways (Sacin), lung clearance index (LCI) and conductive airways (Scond) indexes derived from nitrogen multiple-breath washout test (N2MBW).

DETAILED DESCRIPTION:
Investigational device: PEP-MASK=Positive Expiratory Pressure delivered through a face mask.

Standard Operating Procedures used for evaluating CF lung disease and ventilation inhomogeneity.

Sample size: Based on preliminary data collected on seven subjects who performed nitrogen multiple-breath washout test before and after PEP-MASK, assuming a variation of 20% of Sacin, the study requires a sample size of 18 subjects.

ELIGIBILITY:
Inclusion Criteria:

* CF diagnosis
* Patients hospitalized for a scheduled intravenous antibiotics cycle and regularly followed-up by the CF Centre
* ≥ 15 kilograms
* FEV1 ≥ 40%predicted
* Ability to perform NMBW test
* Ability to perform spirometry
* Willing to adhere to protocol procedures
* Patients in treatment with PEP-MASK

Exclusion Criteria:

* Pulmonary Exacerbation within two last week
* Burkholderia cepacia infection
* Patients in lung transplantation waiting list
* Patients undergoing non invasive mechanical ventilation or oxygen therapy

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 19 (Actual)
Dates: Start 2016-11-21 (Actual); Primary Completion 2022-08 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
Effect of PEP-MASK on ventilation heterogeneity (Sacin) | Right after intervention/sham procedure
  Acinar airways (Sacin) mean difference between treatments

SECONDARY OUTCOMES:
Effect of PEP-MASK on ventilation heterogeneity (Scond) | Right after intervention/sham procedure
  Conductive airways (Scond) mean difference between treatments
Effect of PEP-MASK on ventilation heterogeneity (LCI) | Right after intervention/sham procedure
  Ventilation heterogeneity (LCI) mean difference between treatments
Sputum weight | From the beginning to the end of each intervention/sham procedure
  Sputum weight (grams) will be collected throughout the active or sham interventions
Oxygen saturation | From the beginning to the end of each intervention/sham procedure
  Oxygen saturation (SpO2) will be monitored throughout the active or sham interventions

CONTACTS AND LOCATIONS:
Overall Officials: Carla Colombo, Study Director — Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Locations (2):
- Italy (2):
  - Azienda Ospedaliero-Universitaria Meyer, Florence
  - Centro Regionale di Riferimento Fibrosi Cistica, Milan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Miller MR, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Crapo R, Enright P, van der Grinten CP, Gustafsson P, Jensen R, Johnson DC, MacIntyre N, McKay R, Navajas D, Pedersen OF, Pellegrino R, Viegi G, Wanger J; ATS/ERS Task Force. Standardisation of spirometry. Eur Respir J. 2005 Aug;26(2):319-38. doi: 10.1183/09031936.05.00034805. No abstract available. PMID 16055882
- See also: Standard Operating Procedures LCI — http://www.mbwtraining.com/ECFS_MBW_SOP.pdf